CLINICAL TRIAL: NCT06595121
Title: Comparative Bioavailability Study of Budesonide After Inhalation of Budesonide 1 Mg / 2 Ml Nebuliser Suspension (Test Product 08P1707F0): Administration Without and with Activated Charcoal and Inhalation of Pulmicort® 1.0 Mg / 2 Ml Suspension (Reference Product) in Healthy Subjects
Brief Title: Bioequivalence of IMP 08P1707F0 Relative to Pulmicort® (1.0 Mg/2 Ml Suspension)
Acronym: BUNIPILOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Collaborators: Analytical Clinical Concepts (ACC GmbH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UP-CLI-2022-001
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Budesonide; Charcoal

STUDY DESIGN:
Intervention Model Description: Single dose, randomized, open-label, two-formations, three treatments, four-period, four-sequence, cross-over, at one study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IMP 08P1707F0 without charcoal (Experimental): Budesonide 1mg/2mL nebuliser suspension (08P1707F0) without charcoal
  Interventions: Drug: budesonide
- IMP 08P1707F0 with charcoal (Experimental): Budesonide 1mg/2mL nebuliser suspension (08P1707F0) with charcoal
  Interventions: Drug: budesonide; Other: Activated Charcoal
- Pulmicort 1.0mg/2mL Suspension (Active Comparator): Pulmicort 1.0mg/2mL Suspension (First administration)
  Interventions: Drug: budesonide
- Pulmicort 1.0mg/ML suspension (second administration) (Active Comparator): Pulmicort 1.0mg/ML suspension (second administration)
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — Budesonide 1 mg/2mL nebuliser suspension
  Other Names: IMP 08P1707F0
  Arms: IMP 08P1707F0 with charcoal; IMP 08P1707F0 without charcoal
Drug: budesonide — Pulmicort(r) 1 mg/2mL nebuliser suspension
  Arms: Pulmicort 1.0mg/2mL Suspension; Pulmicort 1.0mg/ML suspension (second administration)
Other: Activated Charcoal — suspension of 10g activated charcoal slurried in 70mL of water
  Arms: IMP 08P1707F0 with charcoal

SUMMARY:
This study aims to demonstrate the bioequivalence between the formulation of Budesonide 1mg/2mL nebuliser suspension (IMP 08P1707F0) relaive to the reference product Pulmicort(r) 1.0mg/2mL suspension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Caucasian, male and female (16 male, 8 female) subjects 18 - 55 years of age
* Body mass index within the range of ≥ 18.5 and ≤ 30.0 kg/m2
* Female subjects of childbearing potential1) agree to undergo pregnancy tests and to use at least an acceptable effective birth control method during the study and until 90 days after study end
* Negative Covid-19 test result
* Findings within the range of clinical acceptability in medical history (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Findings within the range of clinical acceptability in physical examination (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Laboratory values within the normal range (or the clinical investigator considers the deviation to be irrelevant for the purpose of the study)
* Normal Electrocardiograms (ECG) or abnormalities which the clinical investigator does not consider a disqualification for participation in the study
* Normal vital signs (normal blood pressure and heart rate measured under stabilised conditions at screening visit after at least 5 minutes of rest in sitting position: systolic blood pressure 100 - 140 mmHg, diastolic blood pressure 60 - 90 mmHg and heart rate 50 - 100 beats per minute; normal body temperature (Forehead, 35.5 °C - 37.0 °C)) or abnormalities which the clinical investigator does not consider a disqualification for participation in the study (...)

Exclusion Criteria:

* History of hypersensitivity to the study drug or any related drugs or to any of the excipients
* History or presence of any clinically significant cardiovascular, pulmonary, hepatobiliary, renal, haematological, gastrointestinal, endocrinologic, immunologic, dermatologic, neurological, psychiatric, metabolic, musculoskeletal, malignant disease or eye disorders as glaucoma or a family history of glaucoma
* Clinically significant abnormal laboratory values
* Clinically significant ECG findings
* Clinically significant vital signs (...)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Cmax of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
  The maximum concentration in plasma among observed concentrations at pre-specified time points
AUC 0-t of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
  The area under the curve of plasma concentration versus time curve from time O to the last measured concentration

SECONDARY OUTCOMES:
AUC 0-∞ of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
AUC t-∞ of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
AUC O-30 min of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42 and 0.50 hours
t max of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
t 1/2 of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
AUC O-15 min of budesonide for the differents arms | predose, 0.05, .010, 0.17 and 0.25 hours
λz of budesonide for the differents arms | predose, 0.05, .010, 0.17, 0.25, 0.33, 0.42, 0.50, 0.67, 1.00, 1.33, 1.67, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 14.00 and 24.00 hours
  λz Elimination rate constant (calculated by log linear regression of concentrations observed during the terminal phase of elimination)
Incidence of treatment-related adverse events | up to 24 hours
  Occurence and severity of adverse events (serious and non serious adverse events)

CONTACTS AND LOCATIONS:
Locations (1):
- Farmagen IKU Merkezi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After the end of study